CLINICAL TRIAL: NCT01352832
Title: Phase II of The Alabama NSAID Patient Safety Survey: Reducing Disparities in Risk Awareness and Communication
Brief Title: The Alabama NSAIDs Patient Safety Survey, Phase II: Reducing Disparities in Risk Awareness and Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert Weech-Maldonado, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X091029002; 1U18HS016956 (AHRQ)
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Pain Management
Keywords: Chronic NSAID use
MeSH Terms: conditions — Agnosia | interventions — Narrative Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive DVD (Experimental): Patients randomized to this arm will receive a DVD DVD (How To Talk To Your Doctor about NSAIDs, HTTTYD-NSAIDs) that presents culturally appropriate "stories" through which a viewer can learn risk factors for adverse effects related to NSAIDs; and communication behaviors for talking about NSAIDs with their doctor.
  Interventions: Other: Interactive DVD
- Usual Care (Placebo Comparator): Patients randomized to this arm receive their usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Interactive DVD — An interactive DVD (How To Talk To Your Doctor about NSAIDs, HTTTYD-NSAIDs) that presents culturally appropriate "stories" through which a viewer can learn risk factors for adverse effects related to NSAIDs; and communication behaviors for talking about NSAIDs with their doctor.
  Other Names: DVD; Educational Materials; Narrative
  Arms: Interactive DVD
Other: Usual Care — Usual Care
  Other Names: Routine care; Standard Care
  Arms: Usual Care

SUMMARY:
The investigators propose a two-year group randomized trial of physician practices to test the effectiveness of an interactive DVD that presents a culturally appropriate communication training program for patients called "How To Talk To Your Doctor (and Get Your Doctor to Talk to YOU!)" in promoting safe prescription and use of Nonsteroidal anti-inflammatory drugs (NSAIDs) in the outpatient setting (HTTTYD-NSAIDs).

The outcome of interest is safer use of NSAIDs as reported by patients. The aims are to:

Aim 1. Develop an interactive DVD (How To Talk To Your Doctor about NSAIDs, HTTTYD-NSAIDs) that presents culturally appropriate "stories" through which a viewer can learn risk factors for adverse effects related to NSAIDs; and communication behaviors for talking about NSAIDs with their doctor.

Aim 2. Conduct a group-randomized trial to test the following three hypotheses about the effectiveness of the interactive DVD in promoting safer use of NSAIDs:

Hypothesis 1: Intervention group patients will be more likely to report that they had a conversation with their doctor about safe NSAID use than control group patients.

Hypothesis 2: Intervention patients will report significantly fewer risky NSAID ingestion behaviors (e.g., concomitant use of OTC and prescription NSAIDs) than control patients.

Hypothesis 3: There will be no difference in the intervention's effectiveness between African American and White participants.

DETAILED DESCRIPTION:
Nonsteroidal Anti-Inflammatory Drugs (NSAIDs), expose patients to substantial risk of toxicity. Risks are compounded by the fact that patients may frequently take both Over-the-Counter (OTC) and prescription NSAIDs, a fact they often do not report to their physician. Further, our prior work suggests that African American patients may be at greater risk from NSAIDs than whites. While the consequences of unsafe NSAID use are well recognized, effective ways of improving safe use are as yet poorly established. Three findings from medical interaction research suggest that a solution may lie in improving doctor-patient communication. First, patients' communicative behaviors influence those of their doctors. Patients who actively participate by preparing beforehand for the visit, asking questions, and expressing concerns, get more information from their doctor, and in many cases receive more diagnostic and therapeutic action. Second, patients can indeed be easily taught to use active communication behaviors during medical encounters. Third, better communicators have better outcomes.A recent report of the Institute of Medicine (IOM) noted that medication-related injuries are frequent, costly and in many cases preventable and strongly recommended that measures be instituted to strengthen patients' capacities for sound medication self-management and communication.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Chronic NSAIDs (prescribed or recommended by their doctor)
* Seen by a primary care physician

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Physician-Patient Communication | Three months from initial survey
  Patients will report that they had a conversation with their doctor about safe NSAID use

SECONDARY OUTCOMES:
Risk behavior related to NSAID use | Three months post initial survey
  Patients will report risky NSAID ingestion behaviors (e.g., concomitant use of OTC and prescription NSAIDs)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weech-Maldonado, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States